CLINICAL TRIAL: NCT02133612
Title: Phase 2 Study of Adjuvant Chemotherapy With Paclitaxel and Cisplatin in Patients With Advanced Esophageal Cancer
Brief Title: Adjuvant Chemotherapy With Paclitaxel and Cisplatin in Lymph Node-Positive Thoracic Esophageal Squamous Cell Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Jing Huang, M.D, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CH-GI-026
Record Dates: First submitted 2014-05-05; First posted 2014-05-08 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-04

CONDITIONS: Esophageal Cancer
Keywords: esophageal cancer; adjuvant chemotherapy; esophageal surgery; paclitaxel; cisplatin
MeSH Terms: conditions — Esophageal Neoplasms | interventions — TP protocol; Paclitaxel

ARMS (1):
- single arm paclitaxel and cisplatin (Experimental)
  Interventions: Drug: paclitaxel; cisplatin

INTERVENTIONS:
Drug: paclitaxel; cisplatin — The adjuvant chemotherapy regimen consisted of paclitaxel 150mg/m2 intravenously (IV) over 3 hours on day 1, followed by cisplatin 50mg/m2 IV on day 2 every 14 days for 4 to 6 cycles.
  Other Names: Paclitaxel Injection, Beijing Union Pharmaceutical Factory

SUMMARY:
Esophageal cancer is a highly aggressive malignancy with a poor overall outcome.

* Five year survival rate after radical esophagectomy is modest at about 40%.The patients with regional lymph node metastases have worse outcome than those without lymph node metastases.
* No standard postoperative adjuvant chemotherapy has ever been established.

ELIGIBILITY:
Inclusion Criteria:

* ability to give informed consent
* histological proof of thoracic esophageal squamous cell carcinoma with negative proximal and distal margins
* node-positive and pathologic stage M0 .
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Patients were enrolled 4 to 10 weeks after surgery.
* Adequate organ function was required in 2 weeks of registration and was defined as: serum creatinine within normal institutional limit, and creatinine clearance (CrCl) ≥60ml/minute. Aspartate aminotransferase and bilirubin<2 times of upper normal institutional limits.

Exclusion Criteria:

* prior chemotherapy or concurrent radiation therapy before esophagectomy
* R1 or R2 resection
* clinically significant hearing loss or symptomatic peripheral neuropathy during initial examination

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2007-12; Primary Completion 2012-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
3 year overall survival | 5 year

SECONDARY OUTCOMES:
3 year disease-free survival | 5 year

OTHER OUTCOMES:
Number of Participants with Adverse Events | 5 year

CONTACTS AND LOCATIONS:
Overall Officials: Jing Huang, M.D, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Xiao Lv, Beijing, Beijing Municipality, China